CLINICAL TRIAL: NCT06690931
Title: Parkinson's Disease Rehabilitation Using Neurofeedback With Functional Electrical Stimulation and Virtual Reality Feedback for Lower Extremities
Brief Title: Neurofeedback Rehabilitation With FES and VR for PD
Acronym: recoveriX PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: g.tec medical engineering GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1367/2023
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Brain-Computer Interface; Neurofeedback; EEG Feedback; Electrical Stimulation Therapy; Virtual reality
MeSH Terms: conditions — Parkinson Disease | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- BCI group (Experimental): Patients in the BCI group will receive 6 sessions per week during 4 weeks of BCI training with FES and VR feedback (24 sessions in total).
  Interventions: Device: Brain-Computer Interface with FES and VR
- Control group (Sham Comparator): Patients in the control group receive 6 sessions of Motor Imagery + FES + VR therapy per week for 4 weeks (24 sessions in total). Patient in the control group will receive the same instructions as the experimental group.
  Interventions: Device: Motor imagery with Functional Electrical Stimulation and Virtual Reality feedback

INTERVENTIONS:
Device: Brain-Computer Interface with FES and VR — The intervention utilizes the recoveriX PRO system. This is a neurofeedback therapy device that combines Brain-Computer Interface based motor imagery, functional electrical stimulation (FES), and virtual reality (VR). This approach enables participants to engage in motor imagery exercises while receiving real-time feedback based on neural signals.
  Participants will complete a total of 24 recoveriX sessions, scheduled at 6 sessions per week, with each session lasting 1 hour.
  Arms: BCI group
Device: Motor imagery with Functional Electrical Stimulation and Virtual Reality feedback — The participants will train the Motor Imagination (MI) combined with Functional Electrical Stimulation (FES) and Virtual Reality (VR) feedback. Feedback provided to the patients will not be linked to the neural signals.
  The amount of stimulation delivered by the feedback devices (FES and VR) will be similar to the experimental group.
  Arms: Control group

SUMMARY:
recoveriX PRO system is a Brain-Computer Interface (BCI) device that combines Motor Imagination (MI), with Functional Electrical Stimulation (FES) and Virtual Reality (VR) as feedback devices. The user wears an electroencephalography (EEG) cap that registers the neural activity during the mental practice. This system allows the user to control the feedback devices (FES +VR) with the MI.

The goal of this clinical trial is to know the safety and clinical effectiveness of recoveriX-based treatment for improving motor functions in Parkinson's Disease patients. Researchers will compare the functional results obtained by recoveriX system, to the standard treatment based in FES + VR + MI without monitoring the EEG activity.

The questions to answer are:

1. Will Parkinson's patients who undergo recoveriX therapy significantly improve their motor functions?
2. Is the functional improvement achieved with the BCI treatment superior to the standard MI+FES+VR treatment?
3. Is the recoveriX-based therapy as safe as the standard treatment?

Participants will have to perform a complete assessment to evaluate their functionality before and after the intervention (motor skills, walking ability, fatigue, impact of the disease in daily living activities).

Patients in the BCI group will receive 6 sessions per week during 4 weeks of BCI training with FES and VR feedback (24 sessions in total).

Patients in the control group receive 6 sessions of FES + VR therapy per week for 4 weeks (24 sessions in total). Patients in the control group will receive the same instructions as the experimental but will not wear the EEG cap.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD
* HY stage between 1 to 3
* Age between 40 - 80 years old
* Ability to walk independently
* Stable medication usage
* Stable neurological condition
* Able to sign the informed consent.
* Able to follow the study protocol.

Exclusion Criteria:

* Other neurological diseases
* Severe depression
* Uncontrolled diabetes
* Concomitant severe neurologic, cardiopulmonary, or orthopedic disorders
* Debilitating conditions or vision impairment that would impede full participation in the study.
* Unpredictable motor fluctuations
* Pregnant
* Active or passive implanted medical devices such as pacemakers which do not allow the use of FES.
* Implanted metallic fragments in the upper and lower extremities which can limit the use of FES.
* Under the influence of anesthesia or similar medication.
* With fractures or lesions in the upper and lower extremities.
* Inadequate control of a BCI system.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Movement Disorders Society - Unified Parkinson's Disease Rating Scale Section III | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  Motor examination.

SECONDARY OUTCOMES:
Movement Disorders Society - Unified Parkinson's Disease Rating Scale - Sections I, II, IV | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  This scale assesses: Section I - Non-motor activities of daily living; Section II - Motor activities of daily living; Section IV - Motor complications.
Parkinson's Disease Questionnaire | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. It also assesses the impact of Parkinson's on specific dimensions of functioning and wellbeing.
  This scale has 39 items, each item has a 5-point ordinal scoring system. The scale ranges from 0 to 156, where low values are related with better quality of life (QoL) and high values to low QoL.
Modified Fatigue Impact Scale | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  The MFIS is a modified form of the Fatigue Impact Scale (Fisk et al. 1994) based on items derived from interviews with PD patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning.
  Participants rate on a 5-point Likert scale, with 0='Never' to 4='Almost always' their agreement with 21 statements. Total scale (0-84) and subscales for physical (0-36), cognitive (0-40) and psychosocial functioning (0-8). Higher numbers indicate greater fatigue.
Accelerometer Tremor Assessment | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  The tremor will be assessed using a small accelerometer placed at the dorsal side of the wrist and above the medial tibial malleolus. Based on the changes in accelerometry a score is generated quantifying the amount of tremor during rest and movement.
9-Hole Peg Test | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  The test is a standardized, quantitative assessment used to measure finger dexterity.
Timed Up & Go | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  This test measures the time it takes patients to get up from a chair, walk 3 metres, turn around, walk 3 metres back and sit down again.
10 Meter Walk Test | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  The 10MWT assesses walking speed in meters per second over a short distance. Individuals walk 10 meters without assistance and the time is measured for the intermediate 6 meters to allow for acceleration and deceleration.
Freezing Of Gait Questionnaire | All patients will be evaluated two pre-assessments before (at week 0 and week 1) and two post-assessments (at week 5, and week 7) after the intervention.
  The FOGQ assesses Freezing of Gait (FOG) severity unrelated to falls in patients with Parkinson's Disease (PD), FOG frequency, disturbances in gait, and relationship to clinical features conceptually associated with gait and motor aspects (e.g., turning). Currently, FOGQ is the only validated tool available to subjectively assess FOG.
  The scale has 6 items, 4 of these items are related to assess FOG severity and 2 are oriented to assess gait. Each item is assessed from 0 to 4 points. Total score ranges from 0 to 24, and higher scores correspond to more severe FOG.

CONTACTS AND LOCATIONS:
Locations (1):
- g.tec medical engineering GmbH, Schiedlberg, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Castro-Cros M, Sebastian-Romagosa M, Rodriguez-Serrano J, Opisso E, Ochoa M, Ortner R, Guger C, Tost D. Effects of Gamification in BCI Functional Rehabilitation. Front Neurosci. 2020 Aug 21;14:882. doi: 10.3389/fnins.2020.00882. eCollection 2020. PMID 32973435
- [Background] Sieghartsleitner S, Sebastian-Romagosa M, Cho W, Grunwald J, Ortner R, Scharinger J, Kamada K, Guger C. Upper extremity training followed by lower extremity training with a brain-computer interface rehabilitation system. Front Neurosci. 2024 Mar 4;18:1346607. doi: 10.3389/fnins.2024.1346607. eCollection 2024. PMID 38500488
- [Background] Sebastian-Romagosa M, Udina E, Ortner R, Dinares-Ferran J, Cho W, Murovec N, Matencio-Peralba C, Sieghartsleitner S, Allison BZ, Guger C. EEG Biomarkers Related With the Functional State of Stroke Patients. Front Neurosci. 2020 Jul 7;14:582. doi: 10.3389/fnins.2020.00582. eCollection 2020. PMID 32733182
- [Background] Sebastian-Romagosa M, Cho W, Ortner R, Murovec N, Von Oertzen T, Kamada K, Allison BZ, Guger C. Brain Computer Interface Treatment for Motor Rehabilitation of Upper Extremity of Stroke Patients-A Feasibility Study. Front Neurosci. 2020 Oct 21;14:591435. doi: 10.3389/fnins.2020.591435. eCollection 2020. PMID 33192277
- [Background] Sebastian-Romagosa M, Cho W, Ortner R, Sieghartsleitner S, Von Oertzen TJ, Kamada K, Laureys S, Allison BZ, Guger C. Brain-computer interface treatment for gait rehabilitation in stroke patients. Front Neurosci. 2023 Oct 18;17:1256077. doi: 10.3389/fnins.2023.1256077. eCollection 2023. PMID 37920297
- See also: Contact — https://recoverix.com/contact-us/